CLINICAL TRIAL: NCT01452451
Title: A Double-Masked, Randomized, Placebo-Controlled, Multiple Ascending Dose Phase 2 Study to Determine the Tolerability, Pharmacokinetics, and Pharmacodynamics of the GLP 1 Agonist HM11260C in Adult Subjects With Type 2 Diabetes Mellitus on Stable Metformin Monotherapy
Brief Title: Safety, Tolerability, Pharmacokinetics,Pharmacodynamics Study of LAPS-Exendin in Subjects of Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HM-EXC-202
Record Dates: First submitted 2011-10-04; First posted 2011-10-14 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- HM11260C (Active Comparator): HM11260C
  Interventions: Drug: HM11260C

INTERVENTIONS:
Drug: HM11260C — 1, 2, and 4 mg for 8 weekly subcutaneous injections for cohorts W1, W2 and W3. 8, 12 and 16 mg for 3 monthly subcutaneous injections for cohorts M1, M2 and M3
  Other Names: LAPS-Exendin4
  Arms: HM11260C
Drug: Placebo — Placebo for 8 weekly subcutaneous injections for cohorts W1, W2 and W3. Placebo for 3 monthly subcutaneous injections for for cohorts M1, M2 and M3
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of repeated doses of HM11260C when given different regimens in subjects with type 2 diabetes mellitus (T2DM) on stable metformin monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Is male or female and 18 to 65 years of age, inclusive, at screening
* Has a history of T2DM and a stable dose of metformin
* Has HbA1c levels at screening between 7% and 10%

Exclusion Criteria:

* Is pregnant or lactating
* Has type 1 diabetes
* Has a significant change in body weight in the 3 months before screening
* Has a fasting plasma glucose level greater than 240 mg/dL (13.3 mmol/L) at screening
* Has an estimated glomerular filtration rate rate <75 mL/min/1.73 m2 or has ≥75 mL/min/1.73 m2 <estimated glomerular filtration rate <90 mL/min/1.73 m2 with a urine albumin to urine creatinine ratio >30 mg/g.
* Has alanine aminotransferase or aspartate aminotransferase values >2.0 × upper limit of normal or total bilirubin >1.5 × upper limit of normal unless the subject has a known history of Gilbert's syndrome
* Has fasting serum triglycerides >400 mg/dL (>4.52 mmol/L) or >250 mg/dL (>2.85 mmol/L) if not on stable lipid-lowering therapy for at least 4 weeks prior to screening, or has calcitonin ≥50 ng/L. Subjects with a history of Fredrickson's Type I, IV or V hyperlipidemia will be excluded.
* Has any history of GI intolerance, chronic diarrhea, inflammatory bowel disease, partial bypass or gastric banding
* Has any acute illness within 5 days before first study drug administration
* Has elevated amylase, ongoing cholelithiasis, cholecystitis at screening, or history of pancreatitis
* Is a heavy tobacco user(more than 10 cigarettes a day)
* Is a heavy alcohol user
* Has a positive screen for drugs of abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-12; Primary Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events as a measure of safety and tolerability | Up to 106 days
  Number of subjects with adverse events as a measure of safety and tolerability when given different regimens to subjects in T2DM with metformin monotherapy

SECONDARY OUTCOMES:
The pharmacokinetics in repeat-dose | Day 1 up to Day 92
  * Before dosing on the first dosing day (Day 1)
  * After the first dose: 8, 24, 48, 72, 96, 120, and 144 hours after dosing
  * Trough samples (ie, immediately before dosing) will be taken prior to dosing on Days 8, 22, 36, 57, 71, and 85
  * After the last dose (thirteenth dose) at 8, 24, 48, 72, 96, 120, and 144 hours after dosing and 7, 10, 14, 21, 28, and 35 days after dosing to define the elimination period of HM11260C
The pharmacodynamics in repeat-dose | Up to 106 days
  HbA1c, glycosylated albumin, fructosamine, insulin, and fasting glucose: For all cohorts: screening; Day -1; before dosing on Days 29, 57, and 85; and at follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio City, Ohio, United States